CLINICAL TRIAL: NCT03572712
Title: Usefulness of Transcutaneous Capnography to Assess Residual Hypoventilation in Obesity-Hypoventilation Syndrom Treated by Non Invasive Ventilation at Home : a Prospective Study
Acronym: PtcCO2-SOH
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0017
Record Dates: First submitted 2018-06-13; First posted 2018-06-28 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-11

CONDITIONS: Obesity Hypoventilation Syndrome
Keywords: Obesity Hypoventilation Syndrome; Non Invasive Ventilation; Transcutaneous capnography
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Interventional study — every patient will be monitored with a blood gase, a nocturnal oximetry and a transcutaneous capnography

SUMMARY:
Transcutaneous capnography (PtcCo2) recently showed good agreement with blood gases to assess hypercapnia. There is no study that has evaluated the benefit to realise systematically a nocturnal PtcCo2 in the follow-up of home-ventilated patient with obesity hypoventilation syndrome (OHS). The investigators will evaluate the intake bring by nocturnal transcutaneous capnography, compared to nocturnal oximetry and blood gases, to diagnose nocturnal alveolar hypoventilation in a population of patient presenting an OHS, treated by non invasive ventilation (NIV) at home .

DETAILED DESCRIPTION:
Patients will be evaluated once a year in consultation with a blood gases, and then a nocturnal recording at home including a transcutaneous capnography and an oximetry.

Some data will be registered too : cardiovascular and neurological comorbidities, diabetes mellitus, treatment, parameters of the non-invasive ventilation, duration of compliance and apnea-hypopnea index (if available).

The investigators will perform a sequential analysis of nocturnal hypoventilation with first blood gases, then nocturnal oxymetry and to finish nocturnal PtcCo2. It will allow us to determine if PtcCo2 catch up some nocturnal hypoventilation, undetected by the first two exams.

The investigators plan that the study will last 18 months. The analysis will be descriptive. Quantitative variables will be described with mean, standard deviation, minimum, maximum and median. Quantitative variables are presented with number and percentage.

Comparison of blood gas / oximetry association with blood gas / oximetry / transcutaneous capnography using a McNemar test

ELIGIBILITY:
Inclusion Criteria:

* Obesity Hypoventilation Syndrom defined by a diurnal PaCo2> 45 mmHg, in stable conditions, in a patient presenting an obesity (BMI > 30 kg/m²)
* treated by non invasive ventilation since at least 3 weeks, and seen in follow-up consultation

Exclusion Criteria:

* minors
* refusal to participate
* under guardianship or trusteeship
* pregnant woman
* other etiology of hypoventilation : copd, kyphoscoliosis, neuromuscular disorders, diaphragmatic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The pneumology department at Nantes University Hospital follows approximately 400 patients treated by non-invasive ventilation, 250 of whom have SOH The investigators plan to include 150 patients in the active patient line followed at Nantes University Hospital, which will make it possible to obtain the number of patients necessary to obtain satisfactory power while taking into account the fact that a certain number of transcutaneous capnographies will not be conclusive.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
nocturnal hypoventilation | Until 37 days
  Nocturnal PtcCo2 > 49 mmHg more than 10% of sleeping time

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No